CLINICAL TRIAL: NCT00486603
Title: A Phase I/II Trial of Hydroxychloroquine in Conjunction With Radiation Therapy and Concurrent and Adjuvant Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Hydroxychloroquine, Radiation, and Temozolomide Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NABTT-0603; U01CA062475 (NIH); ABTC-0603 (Other: Adult Brain Tumor Consortium); CDR0000549734 (Other: NCI PDQ); NA_00012420 (Other: JHM IRB)
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Hydroxychloroquine; Temozolomide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase 1: RT+TMZ+HCQ 200 mg (Experimental): Phse I: daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT. Starting dose of HCQ is 200mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. After 6 weeks, 4 weeks of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  cohorts of three pts: dose levels: 200, 400, 800mg. NO dose escalation beyond 800mg.
  Other: pharmacological study (PK)
  pts continue on treatment until tumor progression. PKs - correlatives will be collected in Phase 1
  Radiation (RT)
  Interventions: Drug: hydroxychloroquine; Drug: temozolomide; Other: pharmacological study; Radiation: Radiation
- Phase 1: RT+TMZ+HCQ 400 mg (Experimental): Phse I: daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT, 400 mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. After 6 weeks, 4 weeks of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  cohorts of three pts: dose levels: 200, 400, 800mg. NO dose escalation beyond 800mg.
  Other: pharmacological study (PK)
  pts continue on treatment until tumor progression. PKs - correlatives will be collected in Phase 1
  Radiation (RT)
  Interventions: Drug: hydroxychloroquine; Drug: temozolomide; Other: pharmacological study; Radiation: Radiation
- Phase 1: RT+TMZ+HCQ 600 mg (Experimental): Phse I: daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT, 600 mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. After 6 weeks, 4 weeks of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  cohorts of three pts: dose levels: 200, 400, 800mg. NO dose escalation beyond 800mg.
  Other: pharmacological study (PK)
  pts continue on treatment until tumor progression. PKs - correlatives will be collected in Phase 1
  Radiation (RT)
  Interventions: Drug: hydroxychloroquine; Drug: temozolomide; Other: pharmacological study; Radiation: Radiation
- Phase 1: RT+TMZ+HCQ 800 mg (Experimental): Phse I: daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT, 800 mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. After 6 weeks, 4 weeks of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  cohorts of three pts: dose levels: 200, 400, 800mg. NO dose escalation beyond 800mg.
  Other: pharmacological study (PK)
  pts continue on treatment until tumor progression. PKs - correlatives will be collected in Phase 1
  Radiation (RT)
  Interventions: Drug: hydroxychloroquine; Drug: temozolomide; Other: pharmacological study; Radiation: Radiation
- Phase 2: RT + TMZ + HCQ MTD (Experimental): Phse 2: daily hydroxychloroquine (HCQ) (MTD 600mg) on 1st day of RT and concomitant temozolomide for 6wks during RT. After 6 weeks, 4 weeks of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  Other: pharmacological study (PK)
  Pts will continue on treatment until tumor progression. PKs - correlatives will be collected in Phase 2
  Radiation (RT)
  Interventions: Drug: hydroxychloroquine; Drug: temozolomide; Other: pharmacological study; Radiation: Radiation

INTERVENTIONS:
Drug: hydroxychloroquine — see arm description, the first 10 week cycle is call initiation cycle, Post the 10 week cycle of just HCQ, 4 week cycles are called Maintenance Cycles
  Other Names: Plaquenil; HCQ
Drug: temozolomide — TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  Other Names: Temodar; TMZ
Other: pharmacological study — Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Other Names: PK; correlative studies
Radiation: Radiation — Radiation during the first six weeks of treatment Monday-Friday
  Other Names: RT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as hydroxychloroquine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving hydroxychloroquine together with temozolomide and radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of hydroxychloroquine when given together with radiation therapy and temozolomide and to see how well they work in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of hydroxychloroquine when administered in combination with radiotherapy and temozolomide in patients with newly diagnosed glioblastoma multiforme. (Phase I)
* Assess the toxicity of this regimen in these patients. (Phase I)
* Determine the overall survival of patients treated with this regimen. (Phase II)

Secondary

* Assess the frequency of toxicity of this regimen in these patients. (Phase II)
* Evaluate the pharmacokinetics and pharmacodynamics of this regimen in these patients.
* Correlate the average change in autophagic vesicles from baseline with genotype, toxicity, and clinical outcomes.
* Correlate the presence of TP53 and PTEN genes and BECN1 with toxicity and clinical outcomes.

OUTLINE: This is a multicenter, open-label, phase I, dose-escalation study of hydroxychloroquine followed by a phase II study.

* Phase I:

  * Initiation therapy: Patients receive oral temozolomide daily for 6 weeks and undergo conformal or intensity-modulated radiotherapy 5 days a week for 6 weeks. Patients also receive oral hydroxychloroquine daily for 10 weeks beginning concurrently with temozolomide and radiotherapy.

Cohorts of 3-6 patients receive escalating doses of hydroxychloroquine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Maintenance therapy: Beginning 28 days after completion of radiotherapy, patients receive oral temozolomide on days 1-5 and oral hydroxychloroquine on days 1-28. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may then continue to receive hydroxychloroquine alone as above in the absence of disease progression or unacceptable toxicity.

  * Phase II:
* Initiation therapy: Patients receive hydroxychloroquine at the MTD determined in phase I, temozolomide, and radiotherapy as in phase I.
* Maintenance therapy: Patients receive hydroxychloroquine at the MTD determined in phase I and temozolomide as in phase I.

Patients undergo blood and tissue sample collection periodically for pharmacological and correlative studies. Samples are analyzed for the mutational status of TP53 and PTEN genes and copy number of BECN1 via PCR; changes in autophagy protein LC3 via gel electrophoresis; and differences in the formation of LC3-II via immunoblotting.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade IV supratentorial astrocytoma (glioblastoma multiforme)
* Newly diagnosed disease
* Diagnosis must have been made by biopsy or resection ≤ 3 months prior to study entry

INCLUSION CRITERIA:

* Patients must be at least 18 years of age.
* Patients must have histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme), established by biopsy or resection not more than 3 months prior to registration.
* Patients must not have received prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agents (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK or gene therapy), or hormonal therapy for their brain tumor. Glucocorticoid therapy is allowed.
* Patients must have a Karnofsky performance status ≤ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Patients must have the following hematologic, renal and liver function (i.e. absolute neutrophil count > 1500/mm3, platelets > 100,000/mm3, creatinine ≤ 2 times the upper limits of normal (ULN) total bilirubin ≤ 1.5 mg/dl, ALT and AST ≤ 4 times above the upper limits of the institutional norm.
* Patients must be able to provide written informed consent.
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test. The anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant.
* Patients must have a Mini Mental State Exam (MMSE) score of > 15.
* Patients must have tumor tissue form completed and signed by a pathologist. See section 9.5.2 for details.
* Prior concurrent therapy:

  * No prior radiotherapy, chemotherapy, immunotherapy, biologic agents (e.g., immunotoxins, immunoconjugates, antisense agents, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphokine-activated killer cell therapy, or gene therapy), or hormonal therapy for brain tumor
  * No prior polifeprosan 20 with carmustine implant (Gliadel wafer) or GliaSite® brachytherapy
  * No concurrent cytochrome P450 enzyme-inducing anticonvulsant drugs (e.g., phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine)
  * No other concurrent chemotherapeutic or investigational agents for this cancer
  * Concurrent glucocorticoids allowed

EXCLUSION CRITERIA:

* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
* Patients who are pregnant or breast-feeding.
* Patients receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents).
* Patients with a concurrent or prior malignancy, unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Patients who have been free of disease (any prior malignancy) for five years are eligible for this study.
* Patients who have received Gliadel wafers or GliaSite brachytherapy are not eligible.
* Due to risk of disease exacerbation patients with porphyria are not eligible.
* Due to risk of disease exacerbation patients with psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations.
* Patients receiving cytochrome P450 enzyme-inducing anticonvulsant drugs (EIADs) (i.e. phenytoin, carbamazepine, Phenobarbital, primidone or oxcarbazepine).
* Patients with previously documented macular degeneration or diabetic retinopathy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-10-29; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myrna Rosenfeld, MD, PhD, Study Chair — New Approaches to Brain Tumor Therapy/Adult Brain Tumor Consortium
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rosenfeld MR, Ye X, Supko JG, Desideri S, Grossman SA, Brem S, Mikkelson T, Wang D, Chang YC, Hu J, McAfee Q, Fisher J, Troxel AB, Piao S, Heitjan DF, Tan KS, Pontiggia L, O'Dwyer PJ, Davis LE, Amaravadi RK. A phase I/II trial of hydroxychloroquine in conjunction with radiation therapy and concurrent and adjuvant temozolomide in patients with newly diagnosed glioblastoma multiforme. Autophagy. 2014 Aug;10(8):1359-68. doi: 10.4161/auto.28984. Epub 2014 May 20. PMID 24991840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by the Adult Brain Tumor Consortium (ABTC) and patients were recruited from the consortium members outpatient centers.
Groups:
- RT+TMZ+HCQ Phase 1 - 200 mg: Daily Hydroxchloroquine (HCQ) on 1st day of RT and TMZ for 6wks during RT. 200mg. After 6 wks, 4 wkd of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  Phse 2: same schema as above but at the prescribed MTD from Phse 1. PKs - correlatives will be collected in Phse 1 and Phse 2
  hydroxychloroquine: see arm description, the first 10 week cycle is call initiation cycle, Post the 10 week cycle of just HCQ, 4 week cycles are called Maintenance Cycles
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study/Correlative study: Seven samples in total will be collected baseline, initiation cycle -wk3-4, wk9-10, Maintenance Cycle 1Week 4 (C1W4), C2W4, C3W4, C6W4
- RT+TMZ+HCQ Phase 1 - 400 mg: Daily Hydroxchloroquine (HCQ) on 1st day of RT and TMZ for 6wks during RT. 400mg. After 6 wks, 4 wkd of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  Phse 2: same schema as above but at the prescribed MTD from Phse 1. PKs - correlatives will be collected in Phse 1 and Phse 2
  hydroxychloroquine: see arm description, the first 10 week cycle is call initiation cycle, Post the 10 week cycle of just HCQ, 4 week cycles are called Maintenance Cycles
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study/Correlative study: Seven samples in total will be collected baseline, initiation cycle -wk3-4, wk9-10, Maintenance Cycle 1Week 4 (C1W4), C2W4, C3W4, C6W4
- RT+TMZ+HCQ Phase 1 - 600 mg: Daily Hydroxchloroquine (HCQ) on 1st day of RT and TMZ for 6wks during RT. 600mg. After 6 wks, 4 wkd of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  Phse 2: same schema as above but at the prescribed MTD from Phse 1. PKs - correlatives will be collected in Phse 1 and Phse 2
  hydroxychloroquine: see arm description, the first 10 week cycle is call initiation cycle, Post the 10 week cycle of just HCQ, 4 week cycles are called Maintenance Cycles
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study/Correlative study: Seven samples in total will be collected baseline, initiation cycle -wk3-4, wk9-10, Maintenance Cycle 1Week 4 (C1W4), C2W4, C3W4, C6W4
- RT+TMZ+HCQ Phase 1 - 800 mg: Daily Hydroxchloroquine (HCQ) on 1st day of RT and TMZ for 6wks during RT. 800mg. After 6 wks, 4 wkd of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  Phse 2: same schema as above but at the prescribed MTD from Phse 1. PKs - correlatives will be collected in Phse 1 and Phse 2
  hydroxychloroquine: see arm description, the first 10 week cycle is call initiation cycle, Post the 10 week cycle of just HCQ, 4 week cycles are called Maintenance Cycles
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study/Correlative study: Seven samples in total will be collected baseline, initiation cycle -wk3-4, wk9-10, Maintenance Cycle 1Week 4 (C1W4), C2W4, C3W4, C6W4
- RT+TMZ+HCQ Phase 2 - MTD 600 mg: Phse 2: daily hydroxychloroquine (HCQ) (MTD 600mg) on 1st day of RT and concomitant temozolomide for 6wks during RT. After 6 wks, 4 wkd of HCQ alone daily. After 6 wks, 4 wkd of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  Pts will continue on treatment unitl tumor progression. PKs - correlatives will be collected in Phse 2
  Radiation
Period: Overall Study
Arm/Group | RT+TMZ+HCQ Phase 1 - 200 mg | RT+TMZ+HCQ Phase 1 - 400 mg | RT+TMZ+HCQ Phase 1 - 600 mg | RT+TMZ+HCQ Phase 1 - 800 mg | RT+TMZ+HCQ Phase 2 - MTD 600 mg
Started | 3 | 7 | 3 | 3 | 76
Completed | 2 | 6 | 3 | 3 | 76
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for all participants from Phase 1 were analyzed as a group.
Groups:
- RT+TMZ+HCQ Phase 1: Phse I: daily Hydroxychloroquine (HCQ) on 1st day of RT and concomitant TMZ for 6wks during RT. Starting dose of HCQ is 200mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. then every 4 weeks will be cycle of mono therapy of HCQ daily.
  cohorts of three pts: dose levels: 200, 400, 600, 800mg. NO dose escalation beyond 800mg.
  hydroxychloroquine: see arm description, the first 10 week cycle is call initiation cycle, Post the 10 week cycle of just HCQ, 4 week cycles are called Maintenance Cycles
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ TMZ days 1-5 150-20mg/m2 cycles 1-6
  pharmacological study/Correlative study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation 6weeks during initiation cycle Monday - Friday
- RT+TMZ+HCQ Phase 2: Daily hydroxychloroquine (HCQ) (MTD 600mg) on 1st day of RT and temozolomide for 6wks during RT. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ TMZ D1-5 150-20mg/m2 cycles 1-6
  pharmacological study/Correlative study: Seven samples in total collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation 6weeks during initiation cycle Monday - Friday
  Pts will continue on treatment unti/tumor progression.
- Total: Total of all reporting groups
Arm/Group | RT+TMZ+HCQ Phase 1 | RT+TMZ+HCQ Phase 2 | Total
Number analyzed (Participants) | 16 | 76 | 92
Age, Continuous [Median (Full Range); unit: years] | 55 [24 to 69] | 59 [20 to 83] | 58 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 30 | 34
  Male | 12 | 46 | 58
Karnofsky Performance Status [Count of Participants; unit: Participants] — The Karnofsky Performance Score (KPS) measures individual's functional impairment to assess prognosis. Score ranges from 0-100 with a lower score reflecting a worse prognosis. KPS is categorized as follows: 0-40= Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly; 50-70= unable to work; able to live at home and care for most personal needs; varying amount of assistance needed; 80-100= able to carry on normal activity and to work; no special care needed. KPS >=60 is part of eligibility criteria for this study.
  Participants
    100 | 5 | 15 | 20
    90 | 7 | 31 | 38
    80 | 3 | 18 | 21
    70 | 1 | 10 | 11
    60 | 0 | 2 | 2
Surgical Procedure [Count of Participants; unit: Participants]
  Biopsy | 6 | 18 | 24
  Craniotomy | 10 | 58 | 68

OUTCOME MEASURES:

1. Primary Outcome: (Phase I) Maximum Tolerated Dose (MTD) of Hydroxychloroquine (HCQ)
Description: Number of participants who tolerated doses of HCQ without dose limiting toxicity. The highest dose at which participants did not experience dose limiting toxicity was determined as the MTD.
Time Frame: 10 weeks
Population: Cohort 200mg - 3 subjects ; cohort 400mg - 7 subjects; 600mg - 3 subjects; 800mg - 3 subjects
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 - Dose Finding: Phse I: daily Hydroxychloroquine (HCQ) on 1st day of RT and concomitant TMZ for 6wks during RT. Starting dose of HCQ is 200mg. After 6 wks, 4 wkd of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  cohorts of three pts: dose levels: 200, 400, 600mg 800mg. NO dose escalation beyond 800mg.
  temozolomide: TMZ daily 75mg/m2 for 6weeks with RT+HCQ TMZ Maintenance cycle 1-6 150-200mg/m2
  pharmacological study/Correlative study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4 (C2W4), Cycle3 Week4 (C3W4), Cycle6 Week4 (C6W4)
  Radiation 6weeks during initation cycle Monday - Friday
Arm/Group | Phase 1 - Dose Finding
Number analyzed (Participants) | 16
Participants
  200mg: number analyzed (Participants) | 3
  200mg | 3
  400mg: number analyzed (Participants) | 7
  400mg | 7
  600mg: number analyzed (Participants) | 3
  600mg | 3
  800mg: number analyzed (Participants) | 3
  800mg | 0

2. Primary Outcome: (Phase I) Number of Participants Who Experienced Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity defined as: Any DLT must be a toxicity considered at least possibly related to HCQ. DLTs will include any possibly, probably, or definitely HCQ-related Grade 3 or 4 toxicity. Known or reasonably suspected TMZ hematological toxicities will not be considered dose limiting unless the treating physician considers the toxicity to be exacerbated by HCQ. Nonhematological toxicities: Any Grades 3-4 severity (except nausea and vomiting without sufficient antiemetic prophylaxis)
Time Frame: 10 weeks
Population: 1/7 subjects from the 400mg cohort only received 70% of expected dose, therefore this subject was not used for toxicity analysis
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: RT+TMZ+HCQ - 200mg: Daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT. Dose of HCQ is 200mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. -Initiation Phase
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation: Radiation during the first six weeks of treatment Monday-Friday
- Phase 1: RT+TMZ+HCQ - 400mg: Daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT. Dose of HCQ is 400mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. -Initiation Phase
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation: Radiation during the first six weeks of treatment Monday-Friday
- Phase 1: RT+TMZ+HCQ - 600mg: Daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT. Dose of HCQ is 600mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. -Initiation Phase
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation: Radiation during the first six weeks of treatment Monday-Friday
- Phase 1: RT+TMZ+HCQ - 800mg: Daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT. Dose of HCQ is 800mg. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. -Initiation Phase
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation: Radiation during the first six weeks of treatment Monday-Friday
Arm/Group | Phase 1: RT+TMZ+HCQ - 200mg | Phase 1: RT+TMZ+HCQ - 400mg | Phase 1: RT+TMZ+HCQ - 600mg | Phase 1: RT+TMZ+HCQ - 800mg
Number analyzed (Participants) | 3 | 6 | 3 | 3
Participants | 0 | 0 | 0 | 3

3. Primary Outcome: (Phase II) Overall Survival
Description: Number of months alive after end of study participation
Time Frame: 2 years
Population: Only Phase 2 participants were assessed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2: RT + TMZ + HCQ: Daily hydroxychloroquine (HCQ) (MTD 600mg) on 1st day of RT and concomitant temozolomide for 6wks during RT. After 6 weeks, 4 weeks of HCQ alone daily. Complete 10 week cycle -Initiation Phase
  Maintenance cycles 1-6 HCQ daily TMZ D 1-5 150-200mg/m2 every 28 days. Cycles 7+ mono therapy of HCQ daily, every 28 days.
  Other: pharmacological study (PK)
  Pts will continue on treatment until tumor progression.
  PKs - correlatives will be collected in Phase 2
  Radiation (RT)
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation: Radiation during the first six weeks of treatment Monday-Friday
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 76
months | 15.6 [13 to 17]

4. Secondary Outcome: (Phase II) Number of Participants With Grade 3 and 4 Toxicity
Description: Number of participants experiencing Grade 3 and 4 toxicity, as defined by CTCAE v3.0, with a possible, probable or definite relationship to HCQ, TMZ or both
Time Frame: up to 2 years
Population: Only participants from Phase II were assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 76
Participants | 22

5. Secondary Outcome: Pharmocodynamics as Determined by Number of Participants With Autophagy Inhibition
Description: Number of participants with at least 2 peripheral blood mononuclear cell (PBMC) samples that were amenable to electronmicroscopy (EM) who showed an increase of autophagic vacuoles in cells.
Time Frame: up to 9 weeks
Population: Only 40 participants had at least 2 PBMC samples that were amenable to EM, which was required to assess this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 40
Participants
  AV increase | 22
  No AV increase | 18

6. Secondary Outcome: Pharmocodynamics as Determined by Number of Participants With Autophagy Inhibition in Relation to Maximal Concentration (Cmax) of HCQ
Description: Autophagy inhibition is represented by an increase in autophagic vacuoles (AV) in participants with at least 2 peripheral blood mononuclear cell samples that were amenable to EM.
Time Frame: up to 9 weeks
Population: Only participants who had at least 2 PBMC samples that were amenable to EM were assessed for this outcome measure
Measure: Count of Participants; unit: Participants
Groups:
- HCQ Cmax <= 1785 ng/mL: Participants from Phase I and II with a HCQ Cmax <= 1785 ng/mL
  Cmax calculated based on 7 samples collected (baseline, initiation Cycle(C) W3-4, W9-10, Maintenance C1W4, C2W4, C3W4, C6W4)
- HCQ Cmax>1785 ng/mL: Participants from Phase I and II with a HCQ Cmax>1785 ng/mL
  Cmax calculated based on 7 samples collected (baseline, initiation Cycle(C) W3-4, W9-10, Maintenance C1W4, C2W4, C3W4, C6W4)
Arm/Group | HCQ Cmax <= 1785 ng/mL | HCQ Cmax>1785 ng/mL
Number analyzed (Participants) | 22 | 18
Participants
  AV Increase | 10 | 12
  No AV Increase | 12 | 6

7. Secondary Outcome: Pharmacokinetics (PK) of Hydroxychloroquine as Measured by Lag Time (Tlag)
Description: The population model PK parameters do not specifically represent steady-state values, as they were determined from multiple repeated single doses taken from multiple repeated doses taken by the individual patient during their period on the study. To obtain steady state PK parameters, individual estimates were simulated from the population model.
Time Frame: up to 276 days
Population: Only participants from Phase II were assessed for this outcome measure. Data was not collected from 4/76 participants.
Measure: Mean (Full Range); unit: hour
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 72
hour | 1.06 [0.97 to 1.25]

8. Secondary Outcome: PK of Hydroxychloroquine as Measured by Oral Clearance (Liters/Hour) From Central Compartment (CL/F)
Description: as for outcome 7
Time Frame: up to 276 days
Population: Only participants from Phase II were assessed for this outcome measure. Data was not collected from 4/76 participants.
Measure: Mean (Full Range); unit: L/hr
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 72
L/hr | 11.85 [6.41 to 28.18]

9. Secondary Outcome: PK of Hydroxychloroquine as Measured by Volume of Distribution of Central Compartment (V/F)
Description: as for outcome 7
Time Frame: up to 276 days
Population: Only participants from Phase II were assessed for this outcome measure. Data was not collected from 4/76 participants.
Measure: Mean (Full Range); unit: Liters
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 72
Liters | 483.96 [26 to 5483]

10. Secondary Outcome: PK of Hydroxychloroquine as Measured by Distribution Volume of Peripheral Compartment (V2/F)
Description: as for outcome 7
Time Frame: up to 276 days
Population: Only participants from Phase II were assessed for this outcome measure. Data was not collected from 4/76 participants.
Measure: Mean (Full Range); unit: Liters
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 72
Liters | 963 [558 to 2208]

11. Secondary Outcome: PK of Hydroxychloroquine as Measured by First-order Absorption Rate Constant (Ka)
Description: as for outcome 7
Time Frame: up to 276 days
Population: Only participants from Phase II were assessed for this outcome measure. Data was not collected from 4/76 participants.
Measure: Mean (Full Range); unit: hours
Arm/Group | Phase 2: RT + TMZ + HCQ
Number analyzed (Participants) | 72
hours | 0.51 [0.42 to 0.82]

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events not serious are defined as having Grade 1 and Grade 2 severity
Groups:
- Phase 2: RT+TMZ+HCQ - MTD 600mg: Daily hydroxychloroquine (HCQ) on 1st day of RT and concomitant temozolomide for 6wks during RT. Dose of HCQ is 600mg MTD. After 6 wks, 4 wkd of HCQ alone daily. this will complete 10 week cycle. -Initiation Phase
  temozolomide: TMZ daily 75mg/m2 for 6wks with RT+HCQ (TMZ is given only during Initiation cycle)
  pharmacological study: Seven samples in total will be collected baseline, initiation cycle -week3-4, week9-10, Maintenance Cycle 1 Week 4 (C1W4), Cycle2 Week4, Cycle3 Week4, Cycle6 Week4
  Radiation: Radiation during the first six weeks of treatment Monday-Friday
Arm/Group | Phase 1: RT+TMZ+HCQ - 200mg | Phase 1: RT+TMZ+HCQ - 400mg | Phase 1: RT+TMZ+HCQ - 600mg | Phase 1: RT+TMZ+HCQ - 800mg | Phase 2: RT+TMZ+HCQ - MTD 600mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/3 | 0/3 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/3 | 7/7 | 3/3 | 3/3 | 53/76
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 3/3 | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: RT+TMZ+HCQ - 200mg (N=3) | Phase 1: RT+TMZ+HCQ - 400mg (N=7) | Phase 1: RT+TMZ+HCQ - 600mg (N=3) | Phase 1: RT+TMZ+HCQ - 800mg (N=3) | Phase 2: RT+TMZ+HCQ - MTD 600mg (N=76)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 6 (6)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 3 (3)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
decreased depth perception (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — strep bovis (sepsis)
lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 1 (2) | 2 (2) | 8 (10)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9)
white blood cell count decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 8 (8)
platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 9 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: RT+TMZ+HCQ - 200mg (N=3) | Phase 1: RT+TMZ+HCQ - 400mg (N=7) | Phase 1: RT+TMZ+HCQ - 600mg (N=3) | Phase 1: RT+TMZ+HCQ - 800mg (N=3) | Phase 2: RT+TMZ+HCQ - MTD 600mg (N=76)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
mood alteration (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — agitation
alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 14 (14)
alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 6 (6)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
anemia (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 1 (1) | 3 (4) | 37 (38)
anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 15 (15)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (11)
ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 12 (12)
creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 14 (14)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
other (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — general disorder in right eye
fatigue (General disorders) | 0 (0) | 5 (6) | 2 (2) | 2 (2) | 44 (47)
feber (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — 0
hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
other (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — herpes zoster
other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — thrush
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 5 (6) | 1 (1) | 0 (0) | 35 (38)
neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 10 (10)
pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
platelet count decreased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 30 (32)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 9 (10)
serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 13 (13)
weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
white blood cell count decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 2 (2) | 2 (3) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days